CLINICAL TRIAL: NCT07383922
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study Comparing the Efficacy and Safety of FG-M108 Versus Placebo Combined With Standard Chemotherapy in First-line Treatment of Patients With Claudin18.2-Positive Advanced Pancreatic Cancer
Brief Title: A Study of FG-M108+Chemotherapy vs Placebo+Chemotherapy in Claudin18.2-positive Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FutureGen Biopharmaceutical (Beijing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-M108-06
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; First-line treatment; Claudin18.2
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FG-M108 + Chemotherapy (Experimental): FG-M108 300mg/m2 Intravenous drip, day1, every 3 weeks Nab-paclitaxel 125mg/m2 Intravenous drip, day1, 8, every 3 weeks Nab-paclitaxel 125mg/m2 Intravenous drip, day1, 8, every 3 weeks
  Interventions: Drug: FG-M108; Drug: nab paclitaxel; Drug: Gemcitabine (GEM)
- Placebo + Chemotherapy (Active Comparator): Placebo 300mg/m2 Intravenous drip, day1, every 3 weeks Nab-paclitaxel 125mg/m2 Intravenous drip, day1, 8, every 3 weeks Nab-paclitaxel 125mg/m2 Intravenous drip, day1, 8, every 3 weeks
  Interventions: Drug: nab paclitaxel; Drug: Gemcitabine (GEM); Drug: Placebo for FG-M108

INTERVENTIONS:
Drug: FG-M108 — FG-M108 monoclonal antibody will be administered as a minimum 2-hour Intravenous drip.
  Other Names: M108
  Arms: FG-M108 + Chemotherapy
Drug: nab paclitaxel — Nab-paclitaxel will be administered as an Intravenous drip.
  Other Names: Albumin-bound paclitaxel
Drug: Gemcitabine (GEM) — Gemcitabine will be administered as an Intravenous drip.
  Other Names: Gemcitabine Hydrochloride
Drug: Placebo for FG-M108 — Placebo will be administered as an Intravenous drip.
  Arms: Placebo + Chemotherapy

SUMMARY:
Pancreatic cancer, which stands as one of the most lethal malignancies and a leading cause of cancer-related deaths globally, poses a significant challenge to human health worldwide. However, standard chemotherapeutic regimens show limited effectiveness in advanced pancreatic cancer, creating an urgent demand to investigate and develop novel therapeutic targets and combination treatment strategies. The primary objective of this study is to evaluate the efficacy of FG-M108 combined with gemcitabine and nab-paclitaxel (Nab-P+GEM) versus placebo combined with Nab-P+GEM as first-line treatment, as measured by overall survival (OS). This study will also assess safety, tolerability, pharmacokinetics, and the immunogenicity profile of FG-M108 monoclonal antibody, along with its impact on quality of life.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase 3 study designed to evaluate the efficacy and safety of FG-M108 injection combined with Nab-P+GEM versus placebo combined with Nab-P+GEM as first-line treatment in patients with Claudin18.2-positive, unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form, understand the study, are willing to comply with and have the ability to complete all trial procedures;
* Age 18-80 years (inclusive), any gender;
* Histologically or cytologically confirmed unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma, without prior systemic therapy; or for subjects who have received prior neoadjuvant/adjuvant chemotherapy, the time from the last treatment to disease recurrence is >6 months;
* Able to provide archived or fresh pathological tissue for CLDN18.2 testing, with central laboratory testing confirming tumor tissue CLDN18.2 positive (defined as ≥40% of tumor cells with CLDN18.2 membrane staining ≥2+ by central laboratory IHC);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Have at least one measurable tumor lesion according to RECIST 1.1 criteria;
* Expected survival ≥3 months;
* Adequate cardiac, bone marrow, liver, renal function;

Exclusion Criteria:

* Have received a live vaccine within 4 weeks prior to randomization;
* Have received radiotherapy within 2 weeks prior to randomization;
* Have received other anti-tumor drug therapy within 4 weeks or within 5 half-lives of the anti-tumor drug prior to randomization;
* Have undergone major surgery within 4 weeks prior to randomization;
* Have received any clinical study drug treatment within 4 weeks prior to randomization;
* Have previously received any treatment targeting CLDN18.2, such as CLDN18.2 monoclonal/bispecific antibodies, CLDN18.2 CAR-T, or CLDN18.2 ADC;
* Have a history of other (non-study tumor) malignancies within 3 years prior to randomization;
* Have a history of central nervous system metastases and/or carcinomatous meningitis;
* Have adverse reactions from prior treatments that have not recovered to CTCAE v5.0 Grade ≤1 (excluding alopecia and anemia) prior to randomization;
* Have had clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to randomization;
* Have uncontrolled systemic diseases assessed by the investigator, including diabetes, hypertension, pulmonary fibrosis, interstitial lung disease, etc.;
* The investigator judges the subject to have obvious active gastrointestinal bleeding;
* Known history of Hepatitis C or chronic active Hepatitis B;
* Require systemic treatment with corticosteroids (dose >10 mg/day prednisone or equivalent dose of similar drugs) or other immunosuppressants within ≤14 days prior to randomization;
* Any other condition of the subject (e.g., psychological, geographical, or medical condition) that does not permit compliance with the study and follow-up procedures;
* Are pregnant or breastfeeding;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from randomization to deathdue to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months
  PFS is defined as the duration from randomization to the first imaging confirmation of progressive disease per RECIST 1.1 by investigator evaluation or death due to any cause (whichever occurs first).
Objective Response Rate (ORR) | Up to 24 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator evaluation per RECIST 1.1.
Disease control rate (DCR) | Up to 24 months
  DCR is defined as the proportion of participants who have a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as assessed by investigator evaluation per RECIST 1.1.
Duration Of Response (DOR) | Up to 24 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by investigator evaluation per RECIST 1.1 or death due to any cause (whichever occurs first).
Safety assessed by Adverse Events (AEs) | Up to 24 months
  An AE is any adverse medical event that occurs during a clinical study, whether or not related with medicinal product, including signs, symptoms, abnormal laboratory test results and diseases. The incidence and severity of AEs during the clinical study are recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyu Jin, Ph.D, Study Chair — FutureGen Biopharmaceutical (Beijing) Co., Ltd
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China